CLINICAL TRIAL: NCT04523324
Title: Randomized Comparison of the Immunogenicity of Recombinant and Egg-based Influenza Vaccines Among Healthcare Personnel in Israel
Brief Title: Immunogenicity Trial of Recombinant Influenza Vaccine Among HCP in Israel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Abt Associates (Industry); Clalit Research Institute (Other); Soroka University Medical Center (Other); Rabin Medical Center (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 7250; 200-2016-91806 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Influenza
Keywords: Influenza; Healthcare personnel; Immunogenicity; Repeat vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Masking Description: Open-label trial. Eligible HCP who report already having been vaccinated with Vaxigrip at the time they are approached to join the study will be eligible to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RIV4 (Flublok Quadrivalent) (Active Comparator): Flublok® Quadrivalent by Sanofi Pasteur, 45µg of HA per strain
  Interventions: Biological: Flublok™ Quadrivalent by Sanofi, Inc.
- IIV4 (Vaxigrip Quadrivalent) (Active Comparator): VaxigripTetra™ by Sanofi, Inc., 15µg of HA per strain, egg-based
  Interventions: Biological: VaxigripTetra™ by Sanofi, Inc.

INTERVENTIONS:
Biological: Flublok™ Quadrivalent by Sanofi, Inc. — 0.5 mL intramuscular dose of Flublok
  Arms: RIV4 (Flublok Quadrivalent)
Biological: VaxigripTetra™ by Sanofi, Inc. — 0.5 mL intramuscular dose of Vaxigrip
  Arms: IIV4 (Vaxigrip Quadrivalent)

SUMMARY:
This randomized, open-label, active-controlled trial will assess humoral immune responses to a single dose of 2019-20 recombinant hemagglutinin quadrivalent influenza vaccines (RIV4) compared with standard egg-based unadjuvanted quadrivalent influenza vaccines (IIV4) among healthcare personnel (HCP) vaccinated during the previous 2018-19 season with IIV4. The trial will be conducted at two hospital sites in Israel during the 2019-20 influenza season among HCP who were enrolled in the Study of Healthcare Personnel with Influenza and other Respiratory Viruses in Israel (SHIRI).

DETAILED DESCRIPTION:
This is a randomized, open-label study design. Starting in July 2019, approximately 550 to 700 HCP from two hospitals (275-350 per hospital site) in Israel will be enrolled. Following completion of a written consent form, participants will complete an enrollment survey and grant permission for review of information collected during the SHIRI study, including vaccination status and immune response during the SHIRI study years. Participants will complete an enrollment survey and grant permission to include and integrate information collected during the SHIRI study into the current study's data, including health history, influenza vaccination history, and immune response to vaccination during the SHIRI study years. HCP will be randomly assigned 1:1 to receive a single dose of IIV4 licensed in Israel (expected to be Vaxigrip® Quadrivalent, 15µg of HA per strain) or RIV4 (Flublok® Quadrivalent by Sanofi Pasteur, 45µg of HA per strain) during August-October of 2019. Adverse events following vaccination will be monitored and documented. Blood specimens will be collected prior to vaccination and approximately 28 days after to evaluate immune responses to vaccination.

Eligible HCP who were already vaccinated with Vaxigrip, the vaccine that is routinely available in Israel, at the time they are approached to join the study, will be invited to join the study as part of the Vaxigrip arm. Like randomized participants, participants who were vaccinated with Vaxigrip outside the study will complete a written consent form, an enrollment survey and grant permission for review of information collected during the SHIRI study, including vaccination status and immune response during the SHIRI study years. As part of the consent form, participants will record the estimated date that they received the vaccine, and the location, and will authorize study staff to verify the date of current-year Vaxigrip vaccination in the Clalit EMR and with the hospital vaccination staff. Participants will complete an enrollment survey and grant permission to include and integrate information collected during the SHIRI study into the current study's data, including health history, influenza vaccination history, and immune response to vaccination during the SHIRI study years. Blood specimens will be collected approximately 28 days after to evaluate immune responses to vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Current member of Clalit Health Services
* Consent to randomized receipt of influenza vaccination with either RIV4 or IIV4, or, if already vaccinated in the current year outside of the study, consent to receive a post-vaccination blood draw
* Participated in the SHIRI study and received influenza vaccination during the 2018-19 influenza season (Group 1)
* Participated in any year of the SHIRI study, not vaccinated in 2018-2019, but vaccinated in at least one study year (Group 1 supplemental)
* Participated in the SHIRI study during all three years, regardless of vaccination status (Group 1 supplemental)
* Participated in any year of the SHIRI study and had PCR-confirmed influenza virus infection during any of the three study years (Group 2)

Exclusion Criteria:

* Already received an influenza vaccine during the current influenza season
* Not willing or able to get the flu vaccines being used in this study;
* Previous hypersensitivity reaction to the study vaccines, or any vaccine, as reported by the subject
* Received any non-influenza vaccine (e.g., Hepatitis B or other vaccine recommended for HCP) in the 4 weeks prior to the first study visit or plans to receive a vaccine in the 4 weeks following the first study visit
* Currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication), or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive an experimental agent during participation in this study.
* Any condition or employment status that the potential participant or local study site principle investigator (PI) believes may interfere with successful completion of the study prior to December 2019, including being currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Thompson, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center-Beilinson, Petah Tikva

IPD SHARING:
Plan to Share IPD: No
No current plans

REFERENCES:
- [Background] Hirsch A, Katz MA, Laufer Peretz A, Greenberg D, Wendlandt R, Shemer Avni Y, Newes-Adeyi G, Gofer I, Leventer-Roberts M, Davidovitch N, Rosenthal A, Gur-Arie R, Hertz T, Glatman-Freedman A, Monto AS, Azziz-Baumgartner E, Ferdinands JM, Martin ET, Malosh RE, Neyra Quijandria JM, Levine M, Campbell W, Balicer R, Thompson MG; SHIRI workgroup. Study of Healthcare Personnel with Influenza and other Respiratory Viruses in Israel (SHIRI): study protocol. BMC Infect Dis. 2018 Nov 6;18(1):550. doi: 10.1186/s12879-018-3444-7. PMID 30400834
- [Derived] Fowlkes AL, Peretz A, Greenberg D, Hirsch A, Martin ET, Levine MZ, Edwards L, Radke S, Lauring AS, Ferdinands JM, Zhang C, Yoo YM, Dreiher J, Newes-Adeyi G, Azziz-Baumgartner E, Fry AM, Monto AS, Balicer R, Thompson MG, Katz MA. Randomised immunogenicity trial comparing 2019-2020 recombinant and egg-based influenza vaccines among frequently vaccinated healthcare personnel in Israel. Int J Infect Dis. 2024 Dec;149:107260. doi: 10.1016/j.ijid.2024.107260. Epub 2024 Oct 10. PMID 39395753

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 577 HCP were randomly allocated to receive either IIV4 or RIV4. Due to a delay in the delivery of RIV4 vaccines, 67 participants randomized to receive RIV4 had already been vaccinated in the community with IIV4 before the study started. Because they received the same IIV4 brand (Vaxigrip) as the study control vaccine, we allowed them to continue in the study as controls.
Period: Overall Study
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Started | 211 | 366
Completed | 203 | 334
Not Completed | 8 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent) | Total
Number analyzed (Participants) | 203 | 334 | 537
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [37 to 53] | 44 [38 to 57] | 45 [38 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 229 | 362
  Male | 70 | 105 | 175
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Arab | 16 | 22 | 38
  Ethnicity: Jewish, not Ultra-Orthodox | 181 | 305 | 486
  Ethnicity: Jewish, Ultra-Orthodox | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Israel | 203 | 334 | 537

OUTCOME MEASURES:

1. Primary Outcome: Post-vaccination Geometric Mean Titer Against Influenza Virus A/H1N1
Description: The geometric mean of antibody titers following a single dose of RIV4 or IIV4 as measured by hemagglutination inhibition (HI) for influenza virus A/H1N1
Time Frame: Day 28 days after vaccination
Population: Influenza A(H1N1)pdm09 Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
titers | 173.1 [148.5 to 201.7] | 83.9 [74.5 to 94.5]

2. Primary Outcome: Geometric Mean Titer Ratio (GMR) Against Influenza Virus A/H1N1
Description: The ratio of the pre- vs. post-vaccination titer against influenza virus A/H1N1 following a single dose of RIV4 versus IIV4.
Time Frame: 0 to 28 days after vaccination
Population: Influenza A(H1N1)pdm09 Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Mean-Fold Change
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Mean-Fold Change | 4.0 [3.2 to 5.0] | 1.9 [1.6 to 2.2]

3. Primary Outcome: Post-vaccination Geometric Mean Titer Against Egg-grown Influenza Virus A/H3N2
Description: The geometric mean of antibody titers following a single dose of RIV4 or IIV4 as measured by hemagglutination inhibition (HI) for egg-grown influenza virus A/H3N2
Time Frame: Day 28 days after vaccination
Population: Egg-grown influenza A(H3N2) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
titers | 241.9 [211.1 to 277.0] | 175.7 [158.0 to 195.3]

4. Primary Outcome: Geometric Mean Titer Ratio (GMR) Against Egg-grown Influenza Virus A/H3N2
Description: The ratio of the pre- vs. post-vaccination titer against egg-grown influenza virus A/H3N2 following a single dose of RIV4 versus IIV4.
Time Frame: 0 to 28 days after vaccination
Population: egg-grown influenza virus A/H3N2 Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Mean-Fold Change
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Mean-Fold Change | 4.1 [3.4 to 5.0] | 2.4 [2.1 to 2.8]

5. Primary Outcome: Post-vaccination GMT Against Cell-grown Influenza Virus A/H3N2
Description: The geometric mean of antibody titers following a single dose of RIV4 or IIV4 as measured by hemagglutination inhibition (HI) for cell-grown influenza virus A/H3N2
Time Frame: Day 28 days after vaccination
Population: Cell-grown influenza A(H3N2) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Titers | 185.3 [163.4 to 210.1] | 86.7 [78.7 to 95.7]

6. Primary Outcome: Geometric Mean Titer Ratio (GMR) Against Cell-grown Influenza Virus A/H3N2
Description: The ratio of the pre- vs. post-vaccination titer against cell-grown influenza virus A/H3N2 following a single dose of RIV4 versus IIV4.
Time Frame: 0 to 28 days after vaccination
Population: Cell-grown influenza virus A/H3N2 Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Mean-Fold Change
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Mean-Fold Change | 6.1 [5.1 to 7.3] | 2.6 [2.3 to 3.0]

7. Primary Outcome: Post-vaccination Geometric Mean Titer Against Influenza B(Victoria)
Description: The geometric mean of antibody titers following a single dose of RIV4 or IIV4 as measured by hemagglutination inhibition (HI) for Influenza B(Victoria)
Time Frame: Day 28 days after vaccination
Population: Influenza B(Victoria) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
titers | 89.5 [77.7 to 103.2] | 76.0 [68.0 to 84.8]

8. Primary Outcome: Geometric Mean Titer Ratio (GMR) Against Influenza B(Victoria)
Description: The ratio of the pre- vs. post-vaccination titer against Influenza B(Victoria) following a single dose of RIV4 versus IIV4.
Time Frame: 0 to 28 days after vaccination
Population: Influenza B(Victoria) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Mean-Fold Change
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Mean-Fold Change | 1.9 [1.5 to 2.3] | 1.5 [1.3 to 1.7]

9. Primary Outcome: Post-vaccination Geometric Mean Titer Against Influenza B(Yamagata)
Description: The geometric mean of antibody titers following a single dose of RIV4 or IIV4 as measured by hemagglutination inhibition (HI) for Influenza B(Yamagata)
Time Frame: Day 28 days after vaccination
Population: Influenza B(Yamagata) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
titers | 191.1 [165.4 to 220.8] | 108.3 [96.8 to 121.2]

10. Primary Outcome: Geometric Mean Titer Ratio (GMR) Against Influenza B(Yamagata)
Description: The ratio of the pre- vs. post-vaccination titer against Influenza B(Yamagata) following a single dose of RIV4 versus IIV4.
Time Frame: 0 to 28 days after vaccination
Population: Influenza virus B(Yamagata) Hemagglutination Inhibition Assay Outcome
Measure: Geometric Mean (95% Confidence Interval); unit: Mean-Fold Change
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
Number analyzed (Participants) | 203 | 334
Mean-Fold Change | 2.7 [2.2 to 3.4] | 1.5 [1.3 to 1.8]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | RIV4 (Flublok Quadrivalent) | IIV4 (Vaxigrip Quadrivalent)
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/334
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/334
Other Adverse Events (participants affected / at risk) | 0/203 | 0/334

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04523324/Prot_SAP_000.pdf